CLINICAL TRIAL: NCT00124475
Title: Efficacy and Safety of BAL4079 in the Treatment of Severe Refractory Chronic Hand Dermatitis
Brief Title: Efficacy and Safety of a Retinoid for the Treatment of Severe Chronic Hand Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAP00089
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hand Dermatoses
Keywords: Chronic Hand Dermatitis
MeSH Terms: conditions — Hand Dermatoses | interventions — Alitretinoin

INTERVENTIONS:
Drug: alitretinoin

SUMMARY:
The purpose of the study is to determine the therapeutic effect of alitretinoin, a retinoid, on severe, therapy refractory chronic hand dermatitis.

DETAILED DESCRIPTION:
Chronic hand dermatitis (CHaD) is a frequent and distressing disease. Conventional treatments yield mostly unsatisfactory results. In addition, chronic hand dermatitis leads to 2-5% of all applications for permanent disability pensions in some western countries. In a therapeutic dose finding study alitretinoin was clinically effective for patients with moderate to severe chronic hand dermatitis refractory to topical treatment.

Patients with severe refractory CHaD will be allocated either of two active treatments or placebo. The primary objective is to demonstrate the response rate based on physicians global assessment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hand dermatitis, all types including hyperkeratotic, vesicular, fingertip dermatitis
* Lasting for 6 months since initial diagnosis
* Rated severe
* Refractory to standard therapy including non-medicated therapy and avoidance of irritants and allergens
* Refractory to topical steroids

Exclusion Criteria:

* Female patients who are pregnant or want to become pregnant
* Female patients of child bearing potential who cannot use or will not commit to using two effective forms of contraception simultaneously
* Patients whose disease is adequately controlled by standard non-medicated therapy and standard corticosteroid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035
Dates: Start 2004-12; Primary Completion 2006-10 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Physicians global assessment
at week 12 or 24

SECONDARY OUTCOMES:
Response rate per treatment group
Modified total lesion symptom score
Patients global assessment
at week 12 or 24
Time to relapse

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ruzicka, MD, Principal Investigator — University of Düsseldorf, Dermatological Hospital, Germany
Locations (1):
- Thomas Ruzicka, MD, Düsseldorf, Germany

REFERENCES:
- [Background] Ruzicka T, Larsen FG, Galewicz D, Horvath A, Coenraads PJ, Thestrup-Pedersen K, Ortonne JP, Zouboulis CC, Harsch M, Brown TC, Zultak M. Oral alitretinoin (9-cis-retinoic acid) therapy for chronic hand dermatitis in patients refractory to standard therapy: results of a randomized, double-blind, placebo-controlled, multicenter trial. Arch Dermatol. 2004 Dec;140(12):1453-9. doi: 10.1001/archderm.140.12.1453. PMID 15611422